CLINICAL TRIAL: NCT05438563
Title: Focal Prostate Ablation for Low to Intermediate Grade Cancer Utilizing TULSA Profound System
Brief Title: MRI-guided Transurethral Urethral Ultrasound Ablation for the Treatment of Low to Intermediate Grade Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David A. Woodrum, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-001336; NCI-2022-03567 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-05-20; First posted 2022-06-30 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Prostate Carcinoma; Stage I Prostate Cancer AJCC v8; Stage II Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cystoscopy; Biopsy; Glutamate Carboxypeptidase II

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (MRI-guided TULSA) (Experimental): Patients undergo MRI-guided TULSA. Patients may also undergo DRE, cystoscopy, biopsy, bone scan, PSMA PET, and/or mpMRI at screening.
  Interventions: Procedure: MRI-Guided Transurethral Ultrasound Ablation; Other: Questionnaire Administration; Procedure: Digital Rectal Examination; Procedure: Cystoscopy; Procedure: Biopsy; Procedure: Bone Scan; Procedure: PSMA PET Scan; Procedure: Multiparametric Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: MRI-Guided Transurethral Ultrasound Ablation — Undergo MRI-Guided TULSA
  Other Names: MRI-TULSA
Other: Questionnaire Administration — Ancillary studies
Procedure: Digital Rectal Examination — Undergo DRE
  Other Names: DRE
Procedure: Cystoscopy — Undergo cystoscopy
  Other Names: CS
Procedure: Biopsy — Undergo biopsy
  Other Names: Bx; BIOPSY_TYPE
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: PSMA PET Scan — Undergo PSMA PET
  Other Names: Prostate-specific Membrane Antigen PET; PSMA PET; PSMA-Positron emission tomography
Procedure: Multiparametric Magnetic Resonance Imaging — Undergo mpMRI
  Other Names: MP-MRI; mpMRI; Multi-parametric MRI; Multiparametric MRI

SUMMARY:
This clinical trial tests whether the magnetic resonance imaging (MRI)-guided transurethral ultrasound ablation (TULSA) procedure is safe and effective in treating patients with low to intermediate grade prostate cancer. MRI-guided TULSA ablation is a minimally invasive procedure that uses an ultrasound device guided by MRI imaging to deliver high-energy sound waves, producing very high temperature to ablate (destroy) tumor cells in a targeted manner. The MRI-guided TULSA procedure may help patients avoid surgery and help improve prostate cancer patients' quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To perform the TULSA procedure for safety and efficacy outcomes in men aged 45 to 80 years with biopsy-confirmed, National Comprehensive Cancer Network (NCCN) low to intermediate-risk prostate cancer.

SECONDARY OBJECTIVE:

I. To assess patient-reported metrics for quality of life (QOL). II. To assess return to normal activity. III. Compare economic benefit as noted from Expanded Prostate Cancer Index Composite (EPIC) questionnaire.

OUTLINE:

Patients undergo MRI-guided TULSA. Patients may also undergo digital rectal exam (DRE), cystoscopy, biopsy, bone scan, prostate specific membrane antigen (PSMA) positron emission tomography (PET), and/or multiparametric MRI (mpMRI) at screening.

After completion of study treatment, patients are followed at 3, 6, 9, 12, 15, 18, 21 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 45-80 years, with > 10 years life expectancy
* Biopsy-confirmed, NCCN [Gleason Grade (GG) 1, favorable GG 2 and unfavorable GG3] intermediate-risk prostate cancer
* Stage =< T2c, N0, M0
* International Society of Urological Pathology (ISUP) grade group 1, 2, or 3 disease on transrectal ultrasonography (TRUS)-guided biopsy (minimum 8 cores, combination of systematic and MRI fusion-guided) or in-bore biopsy [minimum 3 cores from each Prostate Imaging-Reporting and Data System (PI-RADS) version (v)2 category >= 3 lesion]. Biopsy reported within 12 months of baseline visit, with minimum 6-week interval between biopsy and baseline
* Prostate specific antigen (PSA) =< 20 ng/mL reported within 3 months of baseline
* Treatment naive
* Planned ablation volume < 3.0 cm axial radius from the urethra on mpMRI acquired within 6 months of baseline

Exclusion Criteria:

* Inability to undergo MRI or general anaesthesia
* Suspected tumour > 30 mm from the prostatic urethra or < 14 mm from the prostatic urethra
* Prostate calcifications > 3 mm in maximum extent obstructing ablation of tumor on low-dose pelvic computed tomography (CT)

  * Criteria subject to additional review and approval by sponsor. Alternatively, prospective TRUS to query calcifications or susceptibility-weighted MRI if available may be used to assess calcification. Imaging for calcification screening must be dated within 1 year of baseline visit
* Unresolved urinary tract infection or prostatitis
* History of proctitis, bladder stones, hematuria, history of acute urinary retention, severe neurogenic bladder
* Artificial urinary sphincter, penile implant or intraprostatic implant
* Less than 10 years life expectancy
* Patients who are otherwise not deemed candidates for radical prostatectomy (RP)
* Inability or unwillingness to provide informed consent
* History of anal or rectal fibrosis or stenosis, or urethral stenosis, or other abnormality challenging insertion of devices

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-04-06 (Actual); Primary Completion 2027-03-07 (Estimated); Study Completion 2027-03-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients free from treatment failure | At 24 months post-treatment
  Failure is defined as: delivery of any additional intervention for prostate cancer (local or systemic, including adjuvant therapy); or metastatic disease; or prostate cancer-specific death.
Proportion of patients who maintain both urinary continence and erectile potency | At 12 months
  Continence is defined as 'pad-free' (0 pads/day), and potency is defined as erection firmness sufficient for penetration (Expanded Prostate Cancer Index Composite [EPIC]). Two-sided, 95% Pearson-Clopper confidence interval (CI) will be calculated for each intervention arm separately, and the difference in safety outcomes, along with exact 95% two-sided CI will be calculated.

SECONDARY OUTCOMES:
Biochemical failure | Up to 24 months
  In the absence of a validated threshold for biochemical failure in the setting of ablative therapies, the Phoenix criteria will be adopted for the transurethral ultrasound ablation (TULSA) procedure (nadir + 2 ng/mL). Prostate-specific antigen (PSA) is measured at baseline/procedure, 3, 6, 9, 12, 15, 18, 21, and 24 months. It's measured using Scale Grade Group 1, 2, 3, and 4.
Histologic failure | At 12 months
  The proportion of patients with clinically significant disease on targeted +/- systematic biopsy at 12 months. Clinically significant disease is defined as Gleason grade group 2 or higher. It is measured using scale Grade Group 1, 2, 3, and 4.
Multiparametric magnetic resonance imaging (mpMRI) Prostate Imaging and Reporting and Data System (PI-RADS) version 2 score for each visible lesion | At 24 months post-treatment
  These data will also be collected at 24 months post-initial treatment, for patients who receive repeat TULSA procedure. Findings from for-cause mpMRI will also be captured using Pi-Rads 1-5, 1 being most likely not cancer to 5 being very suspicious.
Total prostate volume | At 24 months post-treatment
  These data will also be collected at 24 months post-initial treatment, for patients who receive repeat TULSA procedure. Findings from for-cause mpMRI will also be captured.
Salvage-free survival | Up to 24 months
  Will be estimated using the Kaplan-Meier method.
Biochemical failure-free survival | Up to 24 months
  Will be estimated using the Kaplan-Meier method.
Histologic failure-free survival | Up to 24 months
  Will be estimated using the Kaplan-Meier method.
Metastasis-free survival | Up to 24 months
  Will be estimated using the Kaplan-Meier method.
Prostate cancer-specific survival | Up to 24 months
  Will be estimated using the Kaplan-Meier method.
Overall survival | Up to 24 months
  Will be estimated using the Kaplan-Meier method.
Change in quality of life | Baseline up to 24 months
  Change from baseline in the EPIC questions 1-7 domains and in the visual analog score will be measured at baseline, 6, 12, 18, and 24 months using Scale Grade Group 1, 2, 3, and 4.
Change in patient-reported genitourinary function | Baseline up to 24 months
  Change from baseline in the EPIC questions 8-21 will be measured using Scale Grade Group 1, 2, 3, and 4.

CONTACTS AND LOCATIONS:
Overall Officials: David A Woodrum, MD, PhD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials